CLINICAL TRIAL: NCT00237653
Title: Relevance of Valganciclovir in Recurrent Bouts of Cryptogenic Inflammatory Bowel Diseases With an Infection by Cytomegalovirus
Brief Title: MICI-CMV:Valganciclovir in Recurrent Bouts of Cryptogenic Inflammatory Bowel Diseases With an Infection by Cytomegalovirus
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: difficulty to include patients
Sponsor: University Hospital, Grenoble (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DCIC 03 21
Record Dates: First submitted 2005-10-11; First posted 2005-10-12 (Estimated); Last update posted 2009-04-03 (Estimated); Status verified 2009-04

CONDITIONS: Cytomegalovirus Infections; Inflammatory Bowel Diseases
Keywords: Valganciclovir; Cytomegalovirus; Cryptogenic inflammatory bowel diseases; Crohn Disease; colitis, ulcerative
MeSH Terms: conditions — Cytomegalovirus Infections; Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative | interventions — Valganciclovir

INTERVENTIONS:
Drug: Valganciclovir

SUMMARY:
The main objective of this study is to demonstrate the relevance of Valganciclovir on recurrent bouts of cryptogenic inflammatory bowel diseases with infection by cytomegalovirus (CMV). The goal is to obtain 90% (for Valganciclovir treated patients) versus 50% (for placebo treated patients) remission at 3 months (including the discontinuation of corticoids or reducing their dose to under 20 mg of prednisone equivalence), without any relapse over the 6 following months.

DETAILED DESCRIPTION:
The cytomegalovirus (CMV) is a DNA virus from the herpes virus family. It is passed on between humans and even if infection is widespread (50 to 80% of people older than 35 are CMV immunoglobulin G positive) it is often asymptomatic for immunocompetent people. However, for immunocompromised people, such an infection takes on particular frequency, expression and seriousness, with a high frequency of attack to the digestive track (CMV colitis).

For immunocompetent people, colitis causes feverish bloody diarrhea associated with abdominal pain. Colitis diagnosis is often late and cases with complications have been reported (digestive bleeding, toxic giant colon and perforation). The endoscopic aspect of colitis is not specific and diagnosis is based on serology, anatomopathology or immunochemistry. Recently, PCR approaches have allowed more sensitive diagnosis.

CMV INVOLVEMENT IN CIBD PHYSIOPATHOLOGY:

Even though CMV involvement in colitis is rare but sure for immunocompetent people, its involvement in CIBD triggering and morbidity has not been solved yet.

Some authors think infection by CMV may act on CIBD as a trigger factor; since 2 cases of CMV colitis coinciding with the onset of a CIBD have been reported. For other authors, infection by CMV acts by direct pathogenicity causing ulcerative lesions of colonic mucosa and just imitates a CIBD without triggering it.

A third hypothesis is that infection by CMV aggravates inflammatory bowel diseases acting as an exacerbating factor.

In all cases, people suffering from CIBD are highly-exposed to infection by CMV due to immunosuppressive treatment (corticoids, cyclosporine, azathioprin, and methotrexate) and the inflammation itself (which is supposed to be a proning factor).

CMV AND POUCHITIS:

Pouchitis is the most common long-term complication after total proctocolectomy. Usually, it can be cured by antibiotic therapy, but in 15% of cases it becomes chronic and turns onto refractory pouchitis which is difficult to cure.

Infection by CMV can imitate a chronic pouchitis from a clinical and endoscopic view. In such cases, it had been shown that Valganciclovir treatment (10mg/kg/day) led to significant improvement over a 21 day treatment period.

CONCLUSION:

Infection by CMV seems to play an important role and has to be taken into account in CIBD physiopathogeny. Probably underestimated since it is not necessarily searched, it could be a triggering factor or a treatment resistance factor. Immunosuppressive drugs used towards recurrent bouts, in particularly cyclosporine, favors viral reactivation. Then, recurrent bouts of CIBD may be complicated by CMV infection. That is why it could be interesting to establish relevance of antiviral treatment on recurrent bouts of CIBD with infection by CMV.

The main objective of this study is to demonstrate relevance of Valganciclovir on recurrent bouts of Cryptogenic Inflammatory Bowel Diseases with infection by Cytomegalovirus. The goal is to obtain 90% (for Valganciclovir treated patients) versus 50% (for placebo treated patients) of remission at 3 months (including the discontinuation of corticoids or reducing their dose to under 20 mg of prednisone equivalence), without any relapse over the 6 following months.

Secondary objectives are:

* Reversal of CMV immunoglobulin G serology and PCR results on colonic biopsies.
* Improvement in appearance of histological lesions
* Reduction in the number of colectomies
* Evaluation of Valganciclovir tolerance and its side effects

ELIGIBILITY:
Inclusion Criteria:

* Patient suffering from Crohn's disease, ulcerative colitis, unclassifiable colitis or pouchitis.
* Disease needing to be treated by corticoids and/or immunosuppressive drugs.
* Infection by cytomegalovirus.
* New attack during the three previous months.

Exclusion Criteria:

* Serious or complicated attack, needing to be operated.
* Patient suffering from a psychiatric disease or is uncooperative.
* Patient suffering from another serious disease.
* Patient already participating in another clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2004-02; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Improvement of Crohns disease activity index score
Diminution or disappearance of gravity criteria
Endoscopy: improvement in appearance of lesions, or healing
Anatomopathology: improvement of histological criteria, or total regression
Anatomopathology: disappearance of viral infection criteria
Virology: reversal of CMV IgG serology and PCR results

CONTACTS AND LOCATIONS:
Overall Officials: Bruno BONAZ, MD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Gastroenterology Department - University Hospital of Grenoble, Grenoble, France

REFERENCES:
- [Background] Orvar K, Murray J, Carmen G, Conklin J. Cytomegalovirus infection associated with onset of inflammatory bowel disease. Dig Dis Sci. 1993 Dec;38(12):2307-10. doi: 10.1007/BF01299914. No abstract available. PMID 8261839
- [Background] Hofkin GA, Ting CD. Case report: recurrence of chronic ulcerative colitis induced by intercurrent cytomegalic virus infection. Md Med J. 1995 Dec;44(12):1047-8. PMID 8544671
- [Background] Rachima C, Maoz E, Apter S, Thaler M, Grossman E, Rosenthal T. Cytomegalovirus infection associated with ulcerative colitis in immunocompetent individuals. Postgrad Med J. 1998 Aug;74(874):486-9. doi: 10.1136/pgmj.74.874.486. PMID 9926125
- [Background] Begos DG, Rappaport R, Jain D. Cytomegalovirus infection masquerading as an ulcerative colitis flare-up: case report and review of the literature. Yale J Biol Med. 1996 Jul-Aug;69(4):323-8. PMID 9273986
- [Background] Vega R, Bertran X, Menacho M, Domenech E, Moreno de Vega V, Hombrados M, Cabre E, Ojanguren I, Gassull MA. Cytomegalovirus infection in patients with inflammatory bowel disease. Am J Gastroenterol. 1999 Apr;94(4):1053-6. doi: 10.1111/j.1572-0241.1999.01013.x. PMID 10201482
- [Background] Kaufman HS, Kahn AC, Iacobuzio-Donahue C, Talamini MA, Lillemoe KD, Hamilton SR. Cytomegaloviral enterocolitis: clinical associations and outcome. Dis Colon Rectum. 1999 Jan;42(1):24-30. doi: 10.1007/BF02235178. PMID 10211516
- [Background] Berk T, Gordon SJ, Choi HY, Cooper HS. Cytomegalovirus infection of the colon: a possible role in exacerbations of inflammatory bowel disease. Am J Gastroenterol. 1985 May;80(5):355-60. PMID 2859801
- [Background] Pfau PR, Lichtenstein GR. Cytomegalovirus infection as a cause of ileoanal pouchitis. Dis Colon Rectum. 2000 Jan;43(1):113-4. doi: 10.1007/BF02237255. No abstract available. PMID 10813135
- [Background] Pfau P, Kochman ML, Furth EE, Lichtenstein GR. Cytomegalovirus colitis complicating ulcerative colitis in the steroid-naive patient. Am J Gastroenterol. 2001 Mar;96(3):895-9. doi: 10.1111/j.1572-0241.2001.03672.x. PMID 11280572
- [Background] Munoz-Juarez M, Pemberton JH, Sandborn WJ, Tremaine WJ, Dozois RR. Misdiagnosis of specific cytomegalovirus infection of the ileoanal pouch as refractory idiopathic chronic pouchitis: report of two cases. Dis Colon Rectum. 1999 Jan;42(1):117-20. doi: 10.1007/BF02235196. PMID 10211531
- [Background] Moonka D, Furth EE, MacDermott RP, Lichtenstein GR. Pouchitis associated with primary cytomegalovirus infection. Am J Gastroenterol. 1998 Feb;93(2):264-6. doi: 10.1111/j.1572-0241.1998.00264.x. PMID 9468256
- [Background] Papadakis KA, Tung JK, Binder SW, Kam LY, Abreu MT, Targan SR, Vasiliauskas EA. Outcome of cytomegalovirus infections in patients with inflammatory bowel disease. Am J Gastroenterol. 2001 Jul;96(7):2137-42. doi: 10.1111/j.1572-0241.2001.03949.x. PMID 11467645
- [Background] Surawicz CM, Myerson D. Self-limited cytomegalovirus colitis in immunocompetent individuals. Gastroenterology. 1988 Jan;94(1):194-9. doi: 10.1016/0016-5085(88)90630-0. PMID 2826283